CLINICAL TRIAL: NCT05937893
Title: Metabolism in the Human Brain Following Consumption of a Keto-ester in Alcohol Use Disorder (AUD) With Proton Magnetic Resonance Spectroscopic Imaging (MRSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000035050; 000 (Other: yctg)
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: BHB Transport; Alcohol Use Disorder
Keywords: BHB; AUD
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol consumer (AC) participants (Other): Adult volunteers who are alcohol consumers drawn from both an outpatient population and recruited heavy drinkers from the community.
  Interventions: Other: Keto-ester followed by Magnetic Resonance Spectroscopic Imaging (MRSI) scans
- Healthy participants (Other): Healthy adult volunteers who are not dependent on alcohol.
  Interventions: Other: Keto-ester followed by Magnetic Resonance Spectroscopic Imaging (MRSI) scans

INTERVENTIONS:
Other: Keto-ester followed by Magnetic Resonance Spectroscopic Imaging (MRSI) scans — Following baseline scans, the participant will orally consume the keto-ester, for subsequent scans which will include repeated BHB MRSI acquisitions to dynamically measure BHB labeling in the brain, followed by a final GABA MRSI acquisition.

SUMMARY:
The objective of this study is to determine whether BHB levels in the brain will be positively associated with alcohol consumption, due to hypothesized enhancement of BHB transport into the brain.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether BHB levels in the brain will be positively associated with alcohol consumption, due to hypothesized enhancement of BHB transport into the brain. Furthermore, BHB levels in identified brain regions will be compared against measures of craving.

The secondary objective of this study is to investigate if GABA levels will be elevated in key brain regions relative to the baseline scan in AC subjects due to preferential BHB metabolism. The goal is to acquire preliminary data to apply for an R01 or equivalent grant submission to pursue this metabolic therapy in greater detail using the state-of-the-art MRSI platform at Yale University to study alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

* For AUD patients: individuals assessed to be with mild to - medium severity according to the DSM-5 criteria.
* For non-dependent heavy at-risk drinkers: must be Individuals who consume more than 14 drinks per week for men or more than 8 drinks per week for women, for at least the last 2 months.
* For healthy controls: must be light drinkers not dependent on alcohol, who consume fewer than 2 drinks per week for at least the last 6 months.
* English speaking
* Can read and understand a study the consent form

Exclusion Criteria:

* Non-English speaking
* Unable to read and understand the consent form
* History of alcohol withdrawal in the last 12 months. This will reduce chances of a volunteer having withdrawal symptoms in the middle of the experiment.
* Participants with a history of psychiatric conditions (that include PTSD, schizophrenia, and bipolar disorders), or a history of neurological conditions
* Women who test positive on a pregnancy test collected on either the screening visit or day of the study.
* Healthy subjects identified with substance use with the exception of tobacco and alcohol will be excluded.
* AC subjects identified with substance use, with the exception of tobacco, alcohol, and mild cannabis use disorder (based on the DSM-5 criteria during the medical history) in the last 6 months, will be excluded.
* Persons unable to refrain from alcohol use for 48 hours and undergo a 10-hour fast prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in BHB levels in the brain | Approximately 90 minutes after Baseline Assessment
  β-hydroxybutyrate blood levels in the brain will be assessed via MRSI.

SECONDARY OUTCOMES:
Change in GABA levels in the brain | Approximately 90 minutes after Baseline Assessment
  GABA levels will be assessed in the brain via MRSI to determine if they are elevated in key brain regions relative to the baseline scan.

CONTACTS AND LOCATIONS:
Overall Officials: Chathura Kumaragamage, PhD, Principal Investigator — Bioimaging SciencesMagnetic Resonance SpectroscopyRadiology & Biomedical Imaging
Locations (1):
- The Anlyan Center (TAC), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study be submitted to the NIMH data archive (NDA) at the NIH.
Time Frame: Following study completion and final funder reporting obligations.
URL: https://nda.nih.gov/